CLINICAL TRIAL: NCT03503136
Title: Nedaplatin Versus Cisplatin and Capecitabine Versus Fluorouracil in Induction Chemotherapy Plus Concurrent Chemoradiotherapy for Locoregionally Advanced NPC： a Phase 3, Multicentre, Non-inferiority, Randomised Factorial Trial
Brief Title: Nedaplatin Versus Cisplatin and Capecitabine Versus Fluorouracil in IC + CCRT for Locoregionally Advanced NPC
Acronym: NX-NPC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Tongji Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Peking University (Other); Air Force Military Medical University, China (Other); Second Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital of Guangdong Pharmaceutical University (Other); First People's Hospital of Foshan (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Cancer Hospital of Guizhou Province (Other); Xiangya Hospital of Central South University (Other); Jilin Provincial Tumor Hospital (Other); Henan Cancer Hospital (Other Government); Hunan Cancer Hospital (Other); Cancer Hospital of Guangxi Medical University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jun Ma, MD, Prof, Sun Yat-sen University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2018-FXY-076
Record Dates: First submitted 2018-04-06; First posted 2018-04-19 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Induction chemotherapy; Concurrent chemoradiotherapy; Nedaplatin; Capecitabine
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; nedaplatin; Capecitabine; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A (TPF+P-RT) (Experimental): Induction docetaxel, cisplatin, and fluorouracil plus concurrent chemoradiotherapy with cisplatin
  Interventions: Drug: docetaxel, cisplatin, and fluorouracil; Drug: cisplatin
- B (TNF+N-RT) (Experimental): Induction docetaxel, nedaplatin, and fluorouracil plus concurrent chemoradiotherapy with nedaplatin
  Interventions: Drug: nedaplatin; Drug: docetaxel, nedaplatin, and fluorouracil
- C (TPX+P-RT) (Experimental): Induction docetaxel, cisplatin, and capecitabine plus concurrent chemoradiotherapy with cisplatin
  Interventions: Drug: cisplatin; Drug: docetaxel, cisplatin, and capecitabine
- D (TNX+N-RT) (Experimental): Induction docetaxel, nedaplatin, and capecitabine plus concurrent chemoradiotherapy with nedaplatin
  Interventions: Drug: docetaxel, nedaplatin, and capecitabine; Drug: nedaplatin

INTERVENTIONS:
Drug: docetaxel, nedaplatin, and capecitabine — Patients receive docetaxel(60 mg/m2 on day 1), nedaplatin (60 mg/m2 on day 1) and capecitabine (625 mg/m2 bid, on Days 1 to 14) every three weeks for three cycles before the radiotherapy.
  Other Names: TNX induction chemotherapy
  Arms: D (TNX+N-RT)
Drug: nedaplatin — Patients receive concurrent nedaplatin (100mg/m2) every three weeks for two cycles during radiotherapy.
  Other Names: N
  Arms: B (TNF+N-RT); D (TNX+N-RT)
Drug: docetaxel, cisplatin, and fluorouracil — Patients receive docetaxel (60mg/m2 on day 1), cisplatin (60mg/m2 on day 1) and fluorouracil (600mg/m2 on Days 1 to 5) every three weeks for three cycles before the radiotherapy.
  Other Names: TPF induction chemotherapy
  Arms: A (TPF+P-RT)
Drug: cisplatin — Patients receive concurrent cisplatin (100mg/m2) every three weeks for two cycles during radiotherapy.
  Other Names: P
  Arms: A (TPF+P-RT); C (TPX+P-RT)
Drug: docetaxel, cisplatin, and capecitabine — Patients receive docetaxel(60 mg/m2 on day 1), cisplatin (60 mg/m2 on day 1) and capecitabine (625 mg/m2 bid, on Days 1 to 14) every three weeks for three cycles before the radiotherapy.
  Other Names: TPX induction chemotherapy
  Arms: C (TPX+P-RT)
Drug: docetaxel, nedaplatin, and fluorouracil — Patients receive docetaxel (60mg/m2 on day 1), nedaplatin (60mg/m2 on day 1) and fluorouracil (600mg/m2 on Days 1 to 5) every three weeks for three cycles before the radiotherapy.
  Other Names: TNF induction chemotherapy
  Arms: B (TNF+N-RT)

SUMMARY:
This is a phase 3, multicentre, non-inferiority, randomised factorial trial. The purpose of this study is to study the efficacy and safety of nedaplatin versus cisplatin, and capecitabine versus fluorouracil in induction docetaxel, cisplatin, and fluorouracil (TPF) plus concurrent chemoradiotherapy with cisplatin (P-RT) in locoregionally advanced nasopharyngeal carcinoma (NPC).

DETAILED DESCRIPTION:
In this study, patients with non-keratinizing NPC and staged III-IVA (except T3-4N0) are randomly assigned to one of the four groups: Group A: TPF+P-RT; Group B: TNF+N-RT; Group C: TPX+P-RT; Group D: TNX+N-RT. In induction chemotherapy, patients will receive docetaxel(60 mg/m2 on day 1), cisplatin or nedaplatin (60 mg/m2 on day 1) and fluorouracil (600 mg/m2 on Days 1 to 5) or capecitabine (625 mg/m2 bid, on Days 1 to 14) every three weeks for three cycles before the radical radiotherapy. Concurrent cisplatin or nedaplatin (100mg/m2 on day 1) was given every three weeks for two cycles during radiotherapy. Patients are stratified according to the treatment centers and stage. The primary endpoint is progression-free survival (PFS). Secondary end points include overall survival (OS), distant failure-free survival (D-FFS), locoregional failure-free survival (LR-FFS), toxic effects, and quality of life (QOL). All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO) histologically type)
* Performance status of Eastern Cooperative Oncology Group (ECOG) grade 0 or 1
* Tumor staged as American Joint Committee on Cance (AJCC) III-IVA (except T3-4N0)
* Adequate marrow: leucocyte count ≥ 4×10^9/L, hemoglobin ≥ 90g/L and platelet count ≥ 100×10^9/L.
* Normal liver and renal function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ ULN; creatinine clearance ≥ 60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.
* Patients who could not tolerate or allergic to capecitabine.
* Illness that would interfere with oral medication, including dysphagia, chronic diarrhea, or ileus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 632 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years
  Progression-free survival is calculated from the date of randomisation to the date of disease progression or death from any cause, whichever is first.

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival is calculated from randomization to death from any cause.
Distant failure-free survival | 3 years
  Distant failure-free survival is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Locoregional failure-free survival | 3 years
  Locoregional failure-free survival is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 (acute toxicity) and RTOG/EORTC (late toxicity) | Up to 3 years
  Incidence of acute and late toxicity
Quality of life (QOL) as assessed by EORTC quality of life questionnaire(QLQ)-C30 | Up to 16 weeks
  QOL was assessed by EORTC QLQ-C30 during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator Principal Investigator, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lai SZ, Li WF, Chen L, Luo W, Chen YY, Liu LZ, Sun Y, Lin AH, Liu MZ, Ma J. How does intensity-modulated radiotherapy versus conventional two-dimensional radiotherapy influence the treatment results in nasopharyngeal carcinoma patients? Int J Radiat Oncol Biol Phys. 2011 Jul 1;80(3):661-8. doi: 10.1016/j.ijrobp.2010.03.024. Epub 2010 Jul 17. PMID 20643517
- [Background] Li WF, Sun Y, Mao YP, Chen L, Chen YY, Chen M, Liu LZ, Lin AH, Li L, Ma J. Proposed lymph node staging system using the International Consensus Guidelines for lymph node levels is predictive for nasopharyngeal carcinoma patients from endemic areas treated with intensity modulated radiation therapy. Int J Radiat Oncol Biol Phys. 2013 Jun 1;86(2):249-56. doi: 10.1016/j.ijrobp.2012.09.003. Epub 2012 Nov 29. PMID 23200171
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Tang LQ, Chen DP, Guo L, Mo HY, Huang Y, Guo SS, Qi B, Tang QN, Wang P, Li XY, Li JB, Liu Q, Gao YH, Xie FY, Liu LT, Li Y, Liu SL, Xie HJ, Liang YJ, Sun XS, Yan JJ, Wu YS, Luo DH, Huang PY, Xiang YQ, Sun R, Chen MY, Lv X, Wang L, Xia WX, Zhao C, Cao KJ, Qian CN, Guo X, Hong MH, Nie ZQ, Chen QY, Mai HQ. Concurrent chemoradiotherapy with nedaplatin versus cisplatin in stage II-IVB nasopharyngeal carcinoma: an open-label, non-inferiority, randomised phase 3 trial. Lancet Oncol. 2018 Apr;19(4):461-473. doi: 10.1016/S1470-2045(18)30104-9. Epub 2018 Feb 28. PMID 29501366
- [Background] Sasaki Y, Tamura T, Eguchi K, Shinkai T, Fujiwara Y, Fukuda M, Ohe Y, Bungo M, Horichi N, Niimi S, et al. Pharmacokinetics of (glycolate-0,0')-diammine platinum (II), a new platinum derivative, in comparison with cisplatin and carboplatin. Cancer Chemother Pharmacol. 1989;23(4):243-6. doi: 10.1007/BF00451649. PMID 2647312
- [Background] Zheng J, Wang G, Yang GY, Wang D, Luo X, Chen C, Zhang Z, Li Q, Xu W, Li Z, Wang D. Induction chemotherapy with nedaplatin with 5-FU followed by intensity-modulated radiotherapy concurrent with chemotherapy for locoregionally advanced nasopharyngeal carcinoma. Jpn J Clin Oncol. 2010 May;40(5):425-31. doi: 10.1093/jjco/hyp183. Epub 2010 Jan 19. PMID 20085903
- [Background] Tang C, Wu F, Wang R, Lu H, Li G, Liu M, Zhu H, Zhu J, Zhang Y, Hu K. Comparison between nedaplatin and cisplatin plus docetaxel combined with intensity-modulated radiotherapy for locoregionally advanced nasopharyngeal carcinoma: a multicenter randomized phase II clinical trial. Am J Cancer Res. 2016 Sep 1;6(9):2064-2075. eCollection 2016. PMID 27725911
- [Background] Lee AW, Ngan RK, Tung SY, Cheng A, Kwong DL, Lu TX, Chan AT, Chan LL, Yiu H, Ng WT, Wong F, Yuen KT, Yau S, Cheung FY, Chan OS, Choi H, Chappell R. Preliminary results of trial NPC-0501 evaluating the therapeutic gain by changing from concurrent-adjuvant to induction-concurrent chemoradiotherapy, changing from fluorouracil to capecitabine, and changing from conventional to accelerated radiotherapy fractionation in patients with locoregionally advanced nasopharyngeal carcinoma. Cancer. 2015 Apr 15;121(8):1328-38. doi: 10.1002/cncr.29208. Epub 2014 Dec 19. PMID 25529384
- [Background] Chen SZ, Chen XM, Ding Y, Wang XC, Zhang F, Mo KL. Combined chemotherapy with cisplatin, docetaxel and capecitabine for metastatic nasopharyngeal carcinoma: a retrospective analysis. Nan Fang Yi Ke Da Xue Xue Bao. 2011 Jun;31(7):1114-8. PMID 21764676